CLINICAL TRIAL: NCT03364660
Title: Task and Physiological Specific Stimulation for Recovery of Autonomic Function, Voluntary Movement, and Standing Using Epidural Stimulation and Training After Severe Spinal Cord Injury
Brief Title: Task-specific Epidural Stimulation Study
Acronym: TSEPI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Louisville (Other)
Collaborators: Christopher Reeve Paralysis Foundation (Other)
Responsible Party: Principal Investigator, Susan Harkema PhD, Professor, University of Louisville
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 16.0179 TS EPI
Record Dates: First submitted 2017-11-16; First posted 2017-12-06 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Spinal Cord Injuries
Keywords: Epidural Stimulation; Spinal Cord Injury; Task-Specific
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (5):
- Acute Epidural Stimulation for Cardiovascular Stability. (Experimental): Participants are assessed both with and without epidural stimulation for cardiovascular stability for persistent hypotension, orthostatic hypotension and autonomic dysreflexia.
  Interventions: Device: Acute epidural stimulation for cardiovascular stability
- Epidural Stimulation for Cardiovascular stability during daily activities (Experimental): Participants assigned to this arm will receive be randomized to receive epidural stimulation specific for cardiovascular function alone or cardiovascular function and standing, or voluntary movement alone or voluntary movement and standing.
  Interventions: Device: Long Term Epidural Stimulation for Cardiovascular Stability
- Voluntary Movement ES + Stand Training (Experimental): Participants assigned to this group will receive epidural stimulation specific for voluntary movement and will also receive stand training.
  Interventions: Device: Participants undergo approximately 4 months of epidural stimulation for voluntary movement plus stand training.
- Cardiovascular ES + Stand Training (Experimental): Participants assigned to this group will receive epidural stimulation specific for cardiovascular function and will also receive stand training.
  Interventions: Device: Long Term Epidural Stimulation for Cardiovascular Stability plus Stand Training
- Epidural Stimulation for Voluntary Movement (Experimental): Participants assigned to this group receive epidural stimulation specifically for voluntary movement.
  Interventions: Device: Participants undergo approximately 4 months of epidural stimulation for voluntary movement.

INTERVENTIONS:
Device: Acute epidural stimulation for cardiovascular stability — Eligible participants will be implanted with 16-electrode epidural array and epidural stimulator in the spinal cord. Participants received mapping for cardiovascular stability.
  Arms: Acute Epidural Stimulation for Cardiovascular Stability.
Device: Long Term Epidural Stimulation for Cardiovascular Stability — Participants undergo approximately 4 months of epidural stimulation for cardiovascular stability, daily.
  Arms: Epidural Stimulation for Cardiovascular stability during daily activities
Device: Participants undergo approximately 4 months of epidural stimulation for voluntary movement. — Participants undergo approximately 4 months of epidural stimulation for voluntary movement 4-7 days weekly.
  Arms: Epidural Stimulation for Voluntary Movement
Device: Long Term Epidural Stimulation for Cardiovascular Stability plus Stand Training — Participants undergo approximately 4 months of epidural stimulation for cardiovascular stability, daily. Standing in a body weight support (BWS) harness on a treadmill or standing in a standing frame with epidural stimulation for standing up to 5 days weekly.
  Arms: Cardiovascular ES + Stand Training
Device: Participants undergo approximately 4 months of epidural stimulation for voluntary movement plus stand training. — Participants undergo approximately 4 months of epidural stimulation for voluntary movement, 4-7 days weekly. Standing in a body weight support (BWS) harness on a treadmill or standing in a standing frame with epidural stimulation for standing up to 5 days weekly. Standing in a body weight support (BWS) harness on a treadmill or standing in a standing frame with epidural stimulation for standing up to 5 days weekly.
  Arms: Voluntary Movement ES + Stand Training

SUMMARY:
The investigators propose to understand the role of lumbosacral spinal cord epidural stimulation (scES) in recovery of autonomic nervous system function, voluntary movement, and standing in individuals with severe spinal cord injury (SCI). Thirty-six individuals with severe SCI who have cardiovascular and respiratory dysfunction and who are unable to voluntarily move the legs or stand will receive scES for cardiovascular function, voluntary movement, or standing with and/or without weight-bearing standing. Training will consist of practicing voluntary movements or standing in the presence of specific scES configurations designed for the voluntary movements of the legs and trunk (Vol-scES), or epidural stimulation configurations specific for standing (Stand-scES). Specific configurations epidural stimulation for cardiovascular function (CV-scES) will be provided during sitting and supine and during maneuvers of orthostatic or cardiovascular stress. The ability to move voluntarily, stand, as well as cardiovascular, respiratory, bladder, bowel and sexual function will be assessed in these individuals with chronic severe spinal cord injury. Quality of life and costs of health care also will be assessed.

DETAILED DESCRIPTION:
Experimental Design

The investigators will enroll, implant and complete the interventions in 36 research participants who have sustained a SCI in the proposed experiments. The investigators anticipate they will need to screen 108 potential research participants to enroll 36 individuals who will complete the study. This sample size will provide sufficient replication per study group (n=4) from which variance and effect size estimates for each study hypothesis can be calculated, and hypothesis tests conducted. The investigators will also select individuals to assure that there are a minimum of 25% (n=9) women to adequately represent the percentage in the SCI population. The investigators will study each cohort of patients comprehensively, and each individual will be allocated to the group interventions based on the method of minimization. Research participants will be randomized into group interventions. This novel approach of conducting repeated experiments with comprehensive assessments in a smaller cohort of patients, rather than a more traditional approach of including a large number of patients and focusing on a single outcome, will advance both clinical and scientific knowledge in this highly complex population. The investigators have found success with the smaller cohort approach because they can employ more rigorous, quantitative and sensitive outcomes that not only inform them about the potential clinical efficacy, but also provide further knowledge of the mechanisms of neural control of movement and other physiological mechanisms related to cardiovascular, respiratory, bladder, bowel and sexual function.

Group A:

* Vol-scES during voluntary leg movement training while sitting or lying supine (A1).
* CV-scES during sitting or lying supine (A2).

Group B:

* Vol-scES during voluntary leg movement training + Stand-ES during stand training (B1).
* CV-ES during sitting or lying supine + Stand-ES during stand training (B2).

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Non-progressive spinal cord injury
* At least 2 years post injury
* Stable medical condition
* Unable to voluntarily move all individual joints of the legs
* Unable to stand independently
* Cardiovascular dysfunction including presence of persistent low blood pressures and/or symptoms of autonomic dysreflexia and/or orthostatic hypotension and/or dysregulation in response to postural changes and/or highly variable blood pressures in a 24 hour period
* Urodynamic dysfunction including dyssynergia and/or inability to void voluntarily and/or low voiding capacity
* Respiratory dysfunction including at least 15% deficit in predicted pulmonary function outcomes

Exclusion Criteria:

* Ventilator dependent
* Untreated painful musculoskeletal dysfunction, fracture or pressure sore
* Untreated psychiatric disorder or ongoing drug abuse
* Cardiovascular, respiratory, bladder, or renal disease unrelated to spinal cord injury
* Bladder botox injections less than 12 months prior to implant
* Colostomy bag, urostomy
* Any implanted pump (i.e., baclofen pump, pain pump, etc)
* Ongoing nicotine use
* Pregnant at the time of enrollment or planning to become pregnant during the time course of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2017-11-08 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Recovery of autonomic control of cardiovascular function as assessed by cardiovascular assessments | up to 20 months
Recovery of voluntary movement as assessed by functional movement assessments | up to 20 months

CONTACTS AND LOCATIONS:
Overall Officials: Susan J Harkema, PhD, Principal Investigator — University of Louisville
Locations (1):
- University of Louisville, Louisville, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data.

REFERENCES:
- [Derived] Angeli CA, Rejc E, Ugiliweneza B, Boakye M, Forrest GF, Brockman K, Vogt J, Logsdon B, Fields K, Harkema SJ. Activity-based recovery training with spinal cord epidural stimulation improves standing performance in cervical spinal cord injury. J Neuroeng Rehabil. 2025 Apr 30;22(1):101. doi: 10.1186/s12984-025-01636-6. PMID 40301929

DOCUMENTS (1):
  • Study Protocol (2019-02-08): https://cdn.clinicaltrials.gov/large-docs/60/NCT03364660/Prot_002.pdf